CLINICAL TRIAL: NCT01440998
Title: Pilot and Translational Study of Dasatinib (NSC#732517) Paclitaxel and Carboplatin in Women With Advanced Stage and Recurrent Endometrial Cancer
Brief Title: Dasatinib, Paclitaxel, and Carboplatin in Treating Patients With Stage III-IV or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03275; NCI-2011-03275 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0252; CDR0000712251; MDA-2011-0252; 8836 (Other: M D Anderson Cancer Center); 8836 (Other: CTEP); P30CA016672 (NIH); P50CA098258 (NIH)
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Mucinous Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Squamous Cell Carcinoma; Endometrial Transitional Cell Carcinoma; Endometrial Undifferentiated Carcinoma; Endometrioid Adenocarcinoma; Recurrent Uterine Corpus Carcinoma; Stage III Uterine Corpus Cancer AJCC v7; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Stage IV Uterine Corpus Cancer AJCC v7; Stage IVA Uterine Corpus Cancer AJCC v7; Stage IVB Uterine Corpus Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Endometrioid | interventions — Carboplatin; Dasatinib; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (dasatinib, paclitaxel, carboplatin) (Experimental): Patients receive induction therapy comprising dasatinib PO QD for 14 days. *Beginning 7 days later, patients receive paclitaxel IV over 3 hours and carboplatin IV on day 1, and dasatinib PO QD on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Dasatinib; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This pilot phase I trial studies how well dasatinib works together with paclitaxel and carboplatin in treating patients with stage III, stage IV, or endometrial cancer that has come back after a period of improvement. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving dasatinib together with paclitaxel and carboplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate pMEK and EphA2 signaling effectors in pre- and post- treatment biopsy tissues from patients with advanced staged measurable primary or recurrent endometrial cancer.

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of adverse events as assessed by Common Terminology Criteria for Adverse Events version 4 (CTCAE v. 4) of dasatinib administered in combination with paclitaxel and carboplatin in patients with advanced staged measurable primary or recurrent endometrial cancer.

II. To record the objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.

III. To describe the progression-free survival and overall survival.

TERTIARY OBJECTIVES:

I. To explore the relationship of micro ribonucleic acid (RNA) 520d-3p (miR520d-3p) and EphA2 in pretreatment biopsies.

II. To evaluate downstream EphA2 signaling effectors, such as CAV-1, pAKT, FAK, paxillin, and p130cas in pre- and post-tissue treatment biopsies.

III. To explore the effect of dasatinib on the expression of other Eph family members such as EphB2 and EphB4.

IV. To quantify circulating tumor cells (CTCs) before and during the individual treatment phases.

OUTLINE:

Patients receive induction therapy comprising dasatinib orally (PO) once daily (QD) for 14 days. *Beginning 7 days later, patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV on day 1, and dasatinib PO QD on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: * Patients who have had prior external-beam pelvic or extended-field pelvic/para-aortic radiation therapy must receive treatment at a reduced dose.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable stage III, stage IV, or recurrent endometrial carcinoma whose potential for cure by surgery or radiation therapy alone is poor
* Patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell, transitional cell carcinoma, and mesonephric carcinoma; uterine carcinosarcoma are not eligible for either COHORT
* All patients must have measurable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT; measurable disease lesions must be amenable to pre- and post- treatment biopsy
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0 to 2
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
* Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to registration
* Patients should have had NO prior chemotherapy agents for advanced or recurrent endometrial cancer; prior chemotherapy administration in conjunction with primary radiation therapy as a radiosensitizer would not exclude a patient from participation in this trial
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcL, equivalent to Common Terminology Criteria (CTCAE version [v]4) grade 1
* Platelets greater than or equal to 100,000/mcL
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTCAE v4 grade 1
* Bilirubin less than or equal to 1.5 x ULN (CTCAE v4 grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 2.5 x ULN (CTCAE v4 grade 1)
* Alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE v4 grade 1)
* Neuropathy (sensory and motor) less than or equal to CTCAE v4 grade 1
* Therapeutic anticoagulation is not contraindicated, but for those patients on therapeutic anticoagulation, alteration in coagulation parameters is expected following initiation of dasatinib; for patients on therapeutic anticoagulation, coagulation parameters should be assessed weekly for the first cycle following initiation of dasatinib, weekly for the first cycle following a dose reduction, and weekly for a minimum of two weeks after stopping dasatinib
* Warfarin is permitted for prophylaxis or treatment of thrombosis; Note: low-molecular weight heparin is permitted provided the patient's prothrombin time (PT)/international normalized ratio (INR) is =< 1.5; for patients on anticoagulation, coagulation parameters should be assessed weekly for the first cycle following initiation of dasatinib, weekly for the first cycle following a dose reduction, and weekly for a minimum of two weeks after stopping dasatinib
* PT such that INR is =< 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) =< 1.5 times the institutional upper limit of normal; patients receiving low-molecular weight heparin for the prevention or treatment of venous thromboembolic disease are eligible if considered clinically stable on their regimen
* Oxygen saturation greater than or equal to 88% on room air (CTCAE 4 < grade 2)
* Patients must have a baseline electrocardiogram (EKG) performed prior to enrolling on study; the EKG must have corrected QT interval (QTc) < 450 msec and must not show evidence of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation must be less than 3 beats in a row)
* Cardiac ejection fraction must be within the institutional range of normal as measured by left ventricular ejection fraction (LVEF) testing; note that baseline and on treatment scans should be performed using the same modality and preferably at the same institution
* Patients must have signed an approved informed consent
* Patients of childbearing potential must have a negative serum pregnancy test prior to study entry and be practicing an effective form of contraception during the study and for at least 6 months after receiving the final treatment of dasatinib
* Patients must be able to swallow whole tablets
* Patients may not have any clinically significant cardiovascular disease including the following:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged QTc >= 480 msec (Fridericia correction)
  * Ejection fraction less than institutional normal
  * Major conduction abnormality (unless a cardiac pacemaker is present)
  * Patients with any cardiopulmonary symptoms of unknown cause (e.g. shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (EKG) to rule out QTc prolongation; the patient may be referred to a cardiologist at the discretion of the principal investigator; patients with underlying cardiopulmonary dysfunction should be excluded from the study

Exclusion Criteria:

* Patients who have isolated recurrences (vaginal, pelvic, or para-aortic) that are amenable to potentially curative treatment with radiation therapy or surgery
* Patients who have had a prior chemotherapy regimen for advanced or metastatic disease are excluded; patients who received adjuvant chemotherapy must be disease-free for at least 6 months
* Patients may have received prior radiation therapy for treatment of endometrial carcinoma; prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, and/or intravaginal brachytherapy, alone or with chemotherapy as a radiation sensitizer; all radiation therapy must be completed at least 4 weeks prior to the first date of study therapy; the prior radiation field, radiation dose, number of fractions and prior radiation start and stop dates must be provided at registration
* Patients who have previously received dasatinib; additionally, patients may not be receiving any other investigational agents; patients may have received prior hormonal therapy for treatment of endometrial carcinoma; all hormonal therapy must be discontinued at least one week prior to the first date of study therapy; patients with known brain metastases should be excluded from this clinical trial
* Patients with serious, non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula or gastrointestinal perforation; patients with an intra-abdominal abscess within 28 days prior to the first date of dasatinib therapy are ineligible
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels; patients who have a history of significant bleeding disorder unrelated to cancer including:

  * Bleeding diathesis, congenital or acquired within one year prior to initiating protocol therapy (e.g. von Willebrand's disease, acquired anti-factor VIII antibodies); significant gastrointestinal (GI) bleeding within three months prior to initiating protocol therapy
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease (treated or untreated), including primary brain tumor, seizures not controlled with standard medical therapy, or any brain metastases
* Patients who have had radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events (CTCAE v4 grade 2 or greater, excluding alopecia) due to agents administered more than 4 weeks earlier
* Patients cannot take St. John's wort or drink grapefruit juice while on study treatment (discontinue St. John wort at least five days before starting dasatinib)
* Patients who have an active pleural or pericardial effusion of any grade
* Patients receiving IV bisphosphonates agree that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia, and may be restarted only if any hypocalcemia has been corrected
* Patients with clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension, defined as systolic > 140 mmHg or diastolic > 90 mm Hg
  * Myocardial infarction or unstable angina within 6 months of the first date of dasatinib therapy
  * New York Heart Association (NYHA) class II or greater congestive heart failure or serious cardiac arrhythmia requiring medication; this would include women with atrial fibrillation, who require rate-controlling medication
  * CTCAE v4 grade 2 or greater peripheral vascular disease
  * History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA), or subarachnoid hemorrhage within six months of the first date of dasatinib therapy
  * Patients with hypokalemia or hypomagnesemia if it cannot be corrected to within normal limits prior to dasatinib treatment
  * Required use of a concomitant medication that can prolong the QT interval
* Patients may not be receiving any prohibited potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors; for these drugs, a washout period of greater than or equal to 7 days is required prior to starting dasatinib treatment
* The concomitant use of histamine (H2) blockers and proton pump inhibitors (PPI's) with dasatinib is not recommended (e.g., famotidine, omeprazole); the use of antacids should be considered in place of H2 blockers or PPIs in patients receiving dasatinib therapy; if antacid therapy is needed, the antacid dose should be administered two hours before or after the dose of dasatinib
* Patients may not be receiving any other investigational agents
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who are pregnant or nursing; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Uterine carcinosarcoma and other sarcomas of the uterus will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09-20 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Change in pMEK expression | Up to 1 year
  Change in pMEK expression will be evaluated.
Change in EphA2 expression | From baseline to up to day 14
  Summary statistics and box plots will be used to describe the distributions of expression of EphA2 and its downstream signaling effectors.

SECONDARY OUTCOMES:
Response rate (complete [CR] or partial response [PR]) according to Response Evaluation Criteria in Solid Tumors version 1.1 | Up to 1 year
  Best overall response will be tabulated. The proportion of patients with CR and with (CR+PR) will be estimated with 95% confidence intervals.
Progression free survival | From start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
  Estimated with the product-limit estimator of Kaplan and Meier and illustrated with Kaplan-Meier plots.
Overall survival | From start of treatment to time of death, assessed up to 1 year
  Estimated with the product-limit estimator of Kaplan and Meier and illustrated with Kaplan-Meier plots.
Numbers of circulating tumor cells (CTCs) | Up to 1 year
  Descriptive statistics will be used to summarize the number of CTCs for patients with each type of response. Estimate the mean number of CTCs for each of these groups with 95% confidence intervals.
Incidence of adverse events as assessed by Common Terminology Criteria for Adverse Events version 4 | Up to 1 year
  Tabulated by grade and relationship to study drug, stratified by whether or not patients had prior pelvic radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coleman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States